CLINICAL TRIAL: NCT05816746
Title: Low-Dose Decitabine Plus Anti-PD-1 Treatment for Relapsed/Refractory Diffuse Large B Cell Lymphoma With Extranodal (Esp. Central Nervous System) Involvement: A PhaseⅡClinical Trial
Brief Title: Decitabine and Anti-PD-1 in R/R DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu Zhao, Chief physician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP in R/R DLBCL-P01
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Large B Cell Lymphoma; Relapse/Recurrence; Extranodal Extension; Central Nervous System Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Extranodal Extension | interventions — Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Decitabine 10mg/d，VD d1-5; PD-1 200mg，d8
  Interventions: Drug: Low-Dose Decitabine plus anti-PD-1

INTERVENTIONS:
Drug: Low-Dose Decitabine plus anti-PD-1 — Decitabine 10mg/d，VD d1-5; PD-1 200mg，d8
  Other Names: DP

SUMMARY:
Patients with relapsed/refractory diffuse large B cell lymphoma with extranodal (esp. central nervous system) involvement treated with Low-Dose Decitabine plus anti-PD-1 regimen. 3 weeks for a cycle, with a total of 2 years or until the disease progress esor unacceptable toxicity occurs, or the patient decides to withdraw from the trial.

DETAILED DESCRIPTION:
To evaluate the effectiveness and safety of patients with relapsed/refractory diffuse large B cell lymphoma with extranodal (esp. central nervous system) involvement treated with Low-Dose Decitabine plus anti-PD-1 regimen. 3 weeks for a cycle, with a total of 2 years or until the disease progress esor unacceptable toxicity occurs, or the patient decides to withdraw from the trial. Enrollment was planned to be completed within 2 years, and all trials were followed up for 12 months after the last enrolled patient completed treatment. All cases will be followed up and the long-term curative effect will be observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* 14-80 years old, male or female;
* Pathologically confirmed relapsed/refractory diffuse large B cell lymphoma with extranodal (central nervous system) involvement;
* Expected survival of more than 3 months;
* AST and ALT ≤ 3.0 ULN; TBIL and CCr ≤ 1.0 ULN;
* Inactive infection and severe mental illness
* ECOG score 0~2
* According to the New York Heart Association (NYHA) cardiac function grading standards, the heart function grading should be grade I or Grade II; Cardiac ejection fraction >50% or not lower than the lower limit of the range of laboratory test values at the study center; No pathological abnormality was found in ECG; There was no clinically significant pericardial effusion or pleural effusion
* The serum pregnancy test of female subjects must be negative
* Signed informed consent

Exclusion Criteria:

* Subjects with any autoimmune disease requiring long-term use of corticosteroids or immunosuppressive drugs or with a history of other tumors;
* Severe uncontrolled medical disease or active infection (including HIV+);
* Active gastrointestinal bleeding or 1 month history of gastrointestinal bleeding;
* Received allogeneic hematopoietic stem cell transplantation within 6 months or are participating in other clinical studies;
* Pregnant or nursing women;
* Subjects who must be forcibly detained for the treatment of mental or physical diseases (e.g. infectious diseases);
* The researcher thinks it is not suitable for this clinical study (such as poor compliance, drug abuse, etc.)
* The situation that the researcher judged was not suitable for inclusion

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1-year
  ORR

SECONDARY OUTCOMES:
Clinical Benefit Rate | 1-year
  The total percentage of subjects who achieved minimal response (MR) or above after treatment
Progression Free Survival | 1-year
  The time interval between first treatment and first recorded progress disease, or death from any cause, the deadline is the date of the last examination
Duration of Remission | 1-year
  The time interval from first recording to disease remission (PR and above criteria) to first recording to PD. For responding subjects with no documented disease progression, the deadline is the date of the last examination
Time to Response | 1-year
  The time interval between subjects first receiving treatment and first recording of disease remission (PR and above)
Overall Survival | 1-year
  The time interval between when the subject first received treatment and when death from any cause was recorded. For subjects whose death is not recorded, the deadline is the most recent point in time at which the subject is still alive

CONTACTS AND LOCATIONS:
Locations (1):
- ChinaPLAGH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Low-Dose Decitabine plus anti-PD-1 treatment for relapsed/refractory diffuse large B cell lymphoma with extranodal (dsp. central nervous system) involvement: A phaseⅡclinical trial

REFERENCES:
- [Result] Nie J, Wang C, Liu Y, Yang Q, Mei Q, Dong L, Li X, Liu J, Ku W, Zhang Y, Chen M, An X, Shi L, Brock MV, Bai J, Han W. Addition of Low-Dose Decitabine to Anti-PD-1 Antibody Camrelizumab in Relapsed/Refractory Classical Hodgkin Lymphoma. J Clin Oncol. 2019 Jun 10;37(17):1479-1489. doi: 10.1200/JCO.18.02151. Epub 2019 Apr 30. PMID 31039052
- [Result] Ansell SM, Minnema MC, Johnson P, Timmerman JM, Armand P, Shipp MA, Rodig SJ, Ligon AH, Roemer MGM, Reddy N, Cohen JB, Assouline S, Poon M, Sharma M, Kato K, Samakoglu S, Sumbul A, Grigg A. Nivolumab for Relapsed/Refractory Diffuse Large B-Cell Lymphoma in Patients Ineligible for or Having Failed Autologous Transplantation: A Single-Arm, Phase II Study. J Clin Oncol. 2019 Feb 20;37(6):481-489. doi: 10.1200/JCO.18.00766. Epub 2019 Jan 8. PMID 30620669
- [Result] Lacy SE, Barrans SL, Beer PA, Painter D, Smith AG, Roman E, Cooke SL, Ruiz C, Glover P, Van Hoppe SJL, Webster N, Campbell PJ, Tooze RM, Patmore R, Burton C, Crouch S, Hodson DJ. Targeted sequencing in DLBCL, molecular subtypes, and outcomes: a Haematological Malignancy Research Network report. Blood. 2020 May 14;135(20):1759-1771. doi: 10.1182/blood.2019003535. PMID 32187361
- [Result] Nayak L, Iwamoto FM, LaCasce A, Mukundan S, Roemer MGM, Chapuy B, Armand P, Rodig SJ, Shipp MA. PD-1 blockade with nivolumab in relapsed/refractory primary central nervous system and testicular lymphoma. Blood. 2017 Jun 8;129(23):3071-3073. doi: 10.1182/blood-2017-01-764209. Epub 2017 Mar 29. PMID 28356247